CLINICAL TRIAL: NCT03594045
Title: A Phase II Study to Evaluate the Efficacy and Safety of Apixaban in the Treatment of Heparin Induced Thrombocytopenia (HIT)
Brief Title: Efficacy and Safety of Apixaban in the Treatment of Heparin Induced Thrombocytopenia (HIT)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of funding by sponsor
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Rachel P. Rosovsky, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-153
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Results first posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-11

CONDITIONS: Heparin-induced Thrombocytopenia; Heparin-induced Thrombocytopenia and Thrombosis
Keywords: Heparin-induced Thrombocytopenia
MeSH Terms: conditions — Thrombosis | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apixaban for HIT (Experimental): Patients with Heparin Induced Thrombocytopenia (HIT) will receive Apixaban, at an initial dose of 10 mg orally twice a day for 7 days followed by 5 mg twice a day for a total of 30 days.
  Interventions: Drug: Apixaban
- Apixaban for HITT (Experimental): Patients with Heparin Induced Thrombocytopenia with Thrombosis (HITT) will receive Apixaban, at an initial dose of 10 mg orally twice a day for 7 days followed by 5 mg twice a day for a total of 3 months.
  Interventions: Drug: Apixaban

INTERVENTIONS:
Drug: Apixaban — Apixaban is an anticoagulant that works by inhibiting the coagulation factor, Factor Xa.

SUMMARY:
This research study is studying a drug as a possible treatment for heparin induced thrombocytopenia (HIT) or Heparin-induced Thrombocytopenia and Thrombosis (HITT).

The drug involved in this study is apixaban.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial.

The FDA (the U.S. Food and Drug Administration) has not approved apixaban as a treatment option for this specific disease but it has been approved for other uses.

HIT and HITT are common and severe complications of heparin therapy. Once patients are diagnosed with either one of these, they are typically switched to a non-heparin anticoagulant (a type of drug that thins your blood). As of now the only drug that is FDA approved for HIT or HITT is argatroban, which is administered continuously through an IV over multiple days and is extremely costly.

In this research study, the investigators are researching the activity and tolerability of apixaban in participants with HIT or HITT. The investigators believe that apixaban will work just as well as argatroban and will be more convenient for this population. The oral route of apixaban allows for the potential outpatient treatment of HIT or HITT which is both convenient and less expensive than treatment with argatroban.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients at MGH and participating Dana Farber/Harvard Cancer Center (DF/HCC) sites.
* Patient must have a diagnosis of HIT or high clinical suspicion of HIT, with a 4 T score of ≥ 5 as calculated by the following criteria:
* Thrombocytopenia

  * Platelet count fall >50 percent and nadir ≥20,000/microL - 2 points
  * Platelet count fall 30 to 50 percent or nadir 10 to 19,000/microL - 1 points
  * Platelet count fall <30 percent or nadir <10,000/microL - 0 points
* Timing of platelet count fall

  * Clear onset between days 5 and 10 or platelet count fall at ≤1 day if prior heparin exposure within the last 30 days - 2 points
  * Consistent with fall at 5 to 10 days but unclear (eg, missing platelet counts), onset after day 10, or fall ≤1 day with prior heparin exposure within 30 to 100 days - 1 point
  * Platelet count fall at <4 days without recent exposure - 0 points
* Thrombosis or other sequelae

  * Confirmed new thrombosis, skin necrosis, or acute systemic reaction after intravenous unfractionated heparin bolus - 2 points
  * Progressive or recurrent thrombosis, non-necrotizing (erythematous) skin lesions, or suspected thrombosis that has not been proven - 1 point
  * None - 0 points
* Other causes for thrombocytopenia

  * None apparent - 2 points
  * Possible - 1 point
  * Definite - 0 points
* Prior to or immediately subsequent to enrollment, the patient must have the diagnosis confirmed by Heparin-PF4 EIA or other accepted confirmatory test to remain on study.
* Patients can be treated with argatroban, bivalirudin or fondaparinux for up to 72 hours prior to enrollment.
* Age 18 years or older.
* ECOG performance status ≤2 (Karnofsky ≥60%)
* Participants must have organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * AST(SGOT) and ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine clearance ≥25 mL/min as was used in the AMPLIFY trial16
* The effects of apixaban on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study entry, for the duration of the study participation, and 4 months after completion of apixaban administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patient requires anticoagulation for a mechanical heart valve.
* Patient requires:

  * anticoagulation for another indication for long-term anticoagulation therapy,
  * dual antiplatelet therapy,
  * treatment with aspirin at a dose of more than 162 mg daily
* Patient has signs of active or ongoing clinically significant hemorrhage.
* Patient has hereditary or acquired coagulopathy or bleeding disorder.
* Patient has a contraindication to apixaban.
* Participants receiving any medications or substances that are inhibitors or inducers of cytochrome P-450 3A4 or p-glycoprotein are ineligible. Because this list of these agents are constantly changing, it is important to regularly consult a frequently-updated list. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Patient has severe renal insufficiency (CrCl <25 ml/min-as used in the AMPLIFY trial)
* Patient has hepatic disease (including Child-Pugh B and C) associated with coagulopathy or clinically relevant bleeding risk.
* Recent (previous seven days), or complicated lumbar puncture or epidural catheter placement or removal.
* Patient has high potential need to undergo a surgical or major invasive procedure in the near future.
* Patient has a history of uncorrected cerebral aneurysm, intracranial tumor or hemorrhagic cerebrovascular accident.
* Patient refuses to receive transfused blood products should this intervention become clinically indicated.
* Patient is taking or has been taking an investigational drug within the previous 30 days prior to enrollment.
* In the judgment of the investigator, any disease or circumstance that would interfere with the objectives of the study.
* Participants with known brain metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to apixaban.
* Uncontrolled intercurrent illness.
* Pregnant women are excluded; breastfeeding should be discontinued if the mother is treated with apixaban.
* Prior treatment with a non-heparin anticoagulant while awaiting study enrollment is not an exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel P Rosovsky, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apixaban for HIT | Apixaban for HITT
Started | 0 | 5
Completed | 0 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No HIT patients were enrolled
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban for HIT | Apixaban for HITT | Total
Number analyzed (Participants) | 0 | 5 | 5
Age, Continuous [Mean (Full Range); unit: years] |  | 68 [54 to 80] | 68 [54 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | 2 | 2
  Male |  | 3 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  | 5 | 5

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of New Symptomatic Thromboembolic Complications (TEC) Within 30 Days of the Initiation of Apixaban
Description: New TEC
Time Frame: 30 days
Population: No HIT patients were enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban for HIT | Apixaban for HITT
Number analyzed (Participants) | 0 | 5
Participants |  | 0

2. Secondary Outcome: Composite Cumulative Incidence of All-cause Mortality, Limb Amputation and New TEC
Description: Composite cumulative incidence
Time Frame: From the start of treatment until 30 days after the end of treatment, up to 60 days total for participants with HIT and up to 120 days total for participants with HITT
Population: No HIT patients were enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban for HIT | Apixaban for HITT
Number analyzed (Participants) | 0 | 5
Participants |  | 0

3. Secondary Outcome: Composite Cumulative Incidence of New TEC and Major Bleeding
Description: Composite cumulative incidence
Time Frame: as for outcome 2
Population: No HIT patients were enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban for HIT | Apixaban for HITT
Number analyzed (Participants) | 0 | 5
Participants |  | 0

4. Secondary Outcome: Cumulative Incidence of Major Bleeding
Description: Major Bleeding
Time Frame: as for outcome 2
Population: No HIT patients were enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban for HIT | Apixaban for HITT
Number analyzed (Participants) | 0 | 5
Participants |  | 0

5. Secondary Outcome: Time to Platelet Recovery
Description: The time to platelet recovery serves as a surrogate index of the activity of apixaban.
Time Frame: From the start of treatment until time of platelet recovery, up to 60 days total for participants with HIT and up to 120 days total for participants with HITT
Population: No HIT patients were enrolled
Measure: Median (Full Range); unit: Days
Arm/Group | Apixaban for HIT | Apixaban for HITT
Number analyzed (Participants) | 0 | 5
Days |  | 2 [2 to 5]

6. Secondary Outcome: Cumulative Incidence of All Cause Mortality
Description: Death due to any cause during treatment or the follow-up period following treatment.
Time Frame: From the start of treatment until the time of death or until 30 days after the end of treatment, up to 60 days total for participants with HIT and up to 120 days total for participants with HITT
Population: No HIT patients were enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban for HIT | Apixaban for HITT
Number analyzed (Participants) | 0 | 5
Participants |  | 0

7. Secondary Outcome: Cumulative Incidence of Limb Amputation
Time Frame: as for outcome 2
Population: No HIT patients were enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban for HIT | Apixaban for HITT
Number analyzed (Participants) | 0 | 5
Participants |  | 0

8. Secondary Outcome: Cumulative Incidence of New Thromboembolic Complications (TEC)
Description: New TEC during the study.
Time Frame: as for outcome 2
Population: No HIT patients were enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Apixaban for HIT | Apixaban for HITT
Number analyzed (Participants) | 0 | 5
Participants |  | 0

ADVERSE EVENTS:
Time Frame: From the start of treatment until 3 days after the last treatment was received, up to approximately 4 months
Description: No HIT patients were enrolled
Arm/Group | Apixaban for HIT | Apixaban for HITT
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/5
Other Adverse Events (participants affected / at risk) | 0/0 | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban for HIT (N=0) | Apixaban for HITT (N=5)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Dizziness (Nervous system disorders) | 0 (0) | 1 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (5)
Fatigue (General disorders) | 0 (0) | 1 (3)
Fever (General disorders) | 0 (0) | 1 (3)
Hematoma (Vascular disorders) | 0 (0) | 1 (3)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (4)
Lung infection (Infections and infestations) | 0 (0) | 1 (6)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (6)
Pain (General disorders) | 0 (0) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Sepsis (Infections and infestations) | 0 (0) | 1 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (6)
Weight loss (Investigations) | 0 (0) | 1 (3)
Wound infection (Infections and infestations) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/45/NCT03594045/Prot_SAP_000.pdf